CLINICAL TRIAL: NCT03509623
Title: Effect of Intravitreal Injection of Aflibercept on Blood Coagulation Parameters in Patients With Age Related Macular Degeneration
Brief Title: Blood Coagulation Parameters in Patients Receiving Intravitreal Aflibercept for Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor in Ophthalmology, University Hospital of Patras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 516/26.7.2017
Record Dates: First submitted 2018-04-04; First posted 2018-04-26 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: neovascular age-related macular degeneration; aflibercept; intravitreal anti-VEGF; coagulation; platelet count; D-Dimer; Fibrinogen
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood coagulation and aflibercept (Experimental): Blood sampling through direct peripheral venous puncture will be collected from treatment naive patients commencing treatment with intravitreal injections of aflibercept for neovascular AMD before the first intravitreal injection of aflibercept and at 7 and 30 days post-injection. Blood coagulation parameters will be evaluated at each timepoint.
  Interventions: Diagnostic Test: Blood sampling through direct peripheral venous puncture

INTERVENTIONS:
Diagnostic Test: Blood sampling through direct peripheral venous puncture — Fasting blood samples will be collected 10-15 minutes before the first intravitreal injection of aflibercept and at 7 and 30 days post-injection using a 19-gauge needle under minimum stasis. Blood coagulation parameters will be evaluated.

SUMMARY:
This study aims to evaluate coagulation parameters in treatment naive patients with neovascular age-related macular degeneration (AMD). Treatment naive patients with neovascular AMD, scheduled to undergo treatment with intravitreal injections of aflibercept will be enrolled in the study. Blood samples will be collected before the first intravitreal injection and at 7 and 30 days after aflibercept administration.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration is one of the leading causes of severe visual loss in the aging population. Intravitreal anti-VEGF agents constitute the mainstay in the treatment of neovascular AMD.

Aflibercept is a recombinant fusion protein targeting vascular endothelial growth factor A(VEGF A) and placenta growth factor (PlGF), developed for intravitreal administration in conditions such as neovascular age related macular degeneration, macular edema due to retinal vein occlusion, diabetic macular edema or myopic choroidal neovascularization. However, treatment with anti-VEGFs like aflibercept, carries a potential risk of arterial thromboembolic events, including stroke and myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* treatment naive patients with neovascular AMD scheduled to undergo treatment with intravitreal aflibercept(IVA) in one eye.

Exclusion Criteria:

* patients under systemic treatment with anti-VEGF agents
* patients under intravitreal anti-VEGF treatment in both eyes
* patients unwilling to return 1 week and 1 month after the first IVA
* patients undergoing dialysis, with chronic liver disease or malignancy, under systemic treatment with nonsteroidal anti-inflammatory drugs or under anticoagulation therapy
* patients with a history of any ATE event during the last 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Change in Platelet count | Samples will be received before the first intravitreal injection, at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in Plasma fibrinogen levels | Samples will be received before the first intravitreal injection, at 7 and 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in Plasma D-dimer levels | Samples will be received before the first intravitreal injection, at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in Activated partial thromboplastin time (aPTT) | Samples will be received before the first intravitreal injection, at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in Prothrombin time (PT) | Samples will be received before the first intravitreal injection, at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in International normalized ratio (INR) | Samples will be received before the first intravitreal injection,at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in Protein S levels | Samples will be received before the first intravitreal injection, at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis
Change in Protein C levels | Samples will be received before the first intravitreal injection, at 7 and at 30 days after aflibercept administration
  Peripheral blood sample analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Georgakopoulos CD, Makri OE, Pallikari A, Kagkelaris K, Plotas P, Grammenou V, Emmanuil A. Effect of intravitreal injection of aflibercept on blood coagulation parameters in patients with age-related macular degeneration. Ther Adv Ophthalmol. 2020 Feb 11;12:2515841420903929. doi: 10.1177/2515841420903929. eCollection 2020 Jan-Dec. PMID 32095777